CLINICAL TRIAL: NCT06924125
Title: Spanish Natural History Study for LAMA2 Muscular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: ASOCIACIÓN IMPÚLSATE PARA LA CURA DE LOS NIÑOS CON DÉFICIT DE MEROSINA (Unknown)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)/433/2021
Record Dates: First submitted 2025-03-07; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: LAMA2-MD (Merosin Deficient Congenital Muscular Dystrophy, MDC1A); Merosin Deficient CMD (Full or Partial); Merosin Deficient Congenital Muscular Dystrophy; Muscular Dystrophies; Cohort Studies
Keywords: Merosin; LAMA2; Laminin; Dystrophy; natural history
MeSH Terms: conditions — Muscular dystrophy congenital, merosin negative; Muscular Dystrophies | interventions — Respiratory Rate; Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma and DNA in selected patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients: Compatible clinical presentation and identification of 2 pathogenic variants in LAMA2, or muscle biopsy with decreased laminin alpha2 protein and at least one pathogenic variant
  Interventions: Diagnostic Test: Motor function scales; Diagnostic Test: MUSCLE ULTRASOUND; Diagnostic Test: Muscle Elastography; Other: Complete physical examination; Other: Ventilatory/ respiratory and other support assessment; Other: Oromotor function and nutrition; Other: Motor Milestone Assessments

INTERVENTIONS:
Diagnostic Test: Motor function scales — Evaluation of patients motor function using motor scales (MFM32, CHOP)
Diagnostic Test: MUSCLE ULTRASOUND — Ultrasound guided evaluation of 28 muscles evaluated accross different body regions, assessed using the Heckmatt gradinf system (semiquantitative scale).
Diagnostic Test: Muscle Elastography — Assess the mechanical properties of muscles, such as stiffness and elasticity.
Other: Complete physical examination — Complete physical evaluations including muscle power and goniometry measurements
Other: Ventilatory/ respiratory and other support assessment — Assessment of ventilatory, respiratory, and other support needs to evaluate the necessity of assistive devices
Other: Oromotor function and nutrition — Assessment of bulbar funcionality: feeding devices, nutritional status.
Other: Motor Milestone Assessments — Motor milestones age of acquisition and loss

SUMMARY:
The objective of this natural history study is to comprehensively characterize the disease progression and clinical features of LAMA2-related dystrophies (LAMA2-RD) in the pediatric population. The study aims to establish a well-defined cohort of patients in Spain, enabling long-term follow-up and facilitating recruitment for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* All patients with compatible clinical presentation and identification of 2 pathogenic variants in LAMA2, or muscle biopsy with decreased laminin alpha2 protein and at least one pathogenic variant
* Signed informed consent by the Legal Authority Responsible and/or assent by the subject (starting from 6 years old)

Ages: 0 Minutes to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with compatible clinical presentation and genetical confirmation LAMA2-RD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Motor function Measurement (MFM32) score | Change from baseline through study completion, an average of 5 years
  Global motor functioning. The items of the MFM are classified in 3 domains: D1: standing and transfers, D2: Axial and proximal motor function, D3: Distal motor function. Higher scored indicate a better outcome. The range of the total score is 0-96. The main point of interest includes the change of MFM score yearly, over a period of 5 years.
Change in Motor Milestones | Change from baseline through study completion, an average of 5 years
  Age at acquisition (yes/no) and loss of all motor functions (ex: Head control, sitting, standing, walking, running, climbing stairs and tip toe walking)
Change in Muscle Echogenicity by Muscle Ultrasound | Change from baseline through study completion, an average of 5 years
  A standardized muscle ultrasound protocol of assessment is performed (whole body). Muscle images are scored using the Heckmatt scale (Score 1-4): Heckmatt grade 1 represents a normal muscle image, Heckmatt grade 2 shows an increased echogenicity without attenuation of the deeper image regions, Heckmatt grade 3 indicates a larger increase in echogenicity with some visible loss of normal muscle architecture, and Heckmatt grade 4 shows a strongly increased echogenicity with complete loss of recognizable muscle architecture.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No